CLINICAL TRIAL: NCT04500860
Title: Low Dose Tadalafil 5mg for Treatment of Female Overactive Bladder Syndrome :6 Months Follow up
Brief Title: Low Dose Tadalafil for Treatment of Female OAB Syndrome: Short Term Follow up.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Urology lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo University
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Female Patients With Overactive Bladder Syndrome or Female Patients With Urgency or Urgency Urinary Incontinence
MeSH Terms: interventions — Tadalafil; Tolterodine Tartrate; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A Tadalafil 5 mg (Active Comparator): 30 patients subjected to Daily dose of tadalafil 5mg
  Interventions: Drug: Low dose tadalafil 5 mg
- Group B Tolterodine (Active Comparator): 30 patients subjected to tolterodine 4 mg daily
  Interventions: Drug: Tolterodine 4 Mg Oral Capsule, Extended Release
- Group C placebo (Placebo Comparator): 30 patients subjected to placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose tadalafil 5 mg — Efficacy of daily low dose tadalafil 5mg for treatment of female overactive bladder syndrome or urgency with or without urgency urinary incontinence
  Arms: Group A Tadalafil 5 mg
Drug: Tolterodine 4 Mg Oral Capsule, Extended Release — To compare efficacy of low dose tadalafil 5 mg to tolterodine 4 mg extended release in treatment of female overactive bladder
  Arms: Group B Tolterodine
Drug: Placebo — Placebo drugs
  Arms: Group C placebo

SUMMARY:
Evaluation of use of low dose tadalafil 5 mg daily for treatment of female OAB syndrome

DETAILED DESCRIPTION:
90 female patients with overactive bladder syndrome divided into 3 groups group A subjected to daily low dose tadalafil 5 mg ,group B subjected to tolterodine and group C to placebo. They are evaluated as using OAB symptoms score for 6 months follow up

ELIGIBILITY:
Inclusion Criteria:

* any female with overactive bladder syndrome, urgency with or without urgency urinary incontinence

Exclusion Criteria:

* Active Urinary tract infection
* neurologic abnormality
* Pure Stress urinary incontinence

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of daily low dose tadalafil 5mg in treatment of female overactive bladder syndrome: 6 months follow up | 6 months
  Evaluation of efficacy of tadalafil 5 mg

CONTACTS AND LOCATIONS:
Locations (1):
- Samer Morsy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided